CLINICAL TRIAL: NCT02485730
Title: Cohort Study for Early Identification of Markers in Cognitively Healthy Family Members of Patients With Alzheimer's Disease
Brief Title: Early Identification of Markers in Alzheimer's Families / ALFA
Acronym: ALFA Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Obra Social La Caixa, Spain (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALFA-FPM-0311
Record Dates: First submitted 2015-06-10; First posted 2015-06-30 (Estimated); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer's Disease
Keywords: Prevention; Cohort Analysis; Healthy Participants
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine and CSF samples collection and analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult children of AD patient: Cognitively healthy adult children of AD patient: First-degree descendant of an AD patient (following diagnosis as define in protocol) from 45 to 64 years old.

SUMMARY:
The ALFA study is a long term, prospective, observational study of AD patients' adult children aimed at studying and characterizing key physio-pathological features of the preclinical phase of AD.

DETAILED DESCRIPTION:
The natural history of AD includes an asymptomatic or preclinical phase characterized by pathological cerebral alterations without any evident symptoms of the disease. The beginning of the preclinical phase can be detected using a series of biological and neuroimaging markers that indicate the presence of Aβ deposition in the brain. A variety of factors such as inflammation, genetic load (e.g., APOE4), diet, cardiovascular risk, sleep disorders and cognitive reserve, produced by endogenous or exogenous factors, vary among individuals and may determine the beginning and evolution of the preclinical phase of the disease. It is possible to identify subclinical, biological, cognitive and neuroimaging changes, in the AD preclinical phase. The longitudinal study of intra-individual changes will be more sensitive than cross-sectional inter-individual studies to detect the cognitive evolution during the AD preclinical phase. Similarly, it would be possible to identify factors in subjects at the preclinical phase that will influence their evolution to the clinical stage of the disease.

The study will start with a screening of 3.000 recruited volunteers (NCT01835717) complying as much as possible with study selection criteria and perfectly aware of the study needs.

The selected 400 participants fulfilling the inclusion criteria will undergo detailed phenotyping consisting in: clinical history, AD family history, full cognitive evaluation, cognitive reserve determination, CSF sample collection, blood and urine sample collection, neuroimaging (MRI), quality of life and habits of life questionnaires (physical activity, diet, sleeping habits, social activity, toxics habits, pollution exposure).

The longitudinal study will consist in a every 3-year follow-up visit in which the participant will undergo a review of the clinical history data, a full cognitive evaluation, neuroimaging (MRI), samples collection (blood, urine, CSF) and update of the life habits changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult children of AD patient: First-degree descendant of an AD patient (following diagnosis as define in protocol).
* Age: 45 to 64 years old.
* Long-term commitment to the study: baseline and follow-up visits. Potential participants have to agree to undergo to all the procedures described in the protocol.

Exclusion Criteria:

* Cognitive impairment: to be included the participant must show no signs of objective cognitive impairment.
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol.
* Illiteracy or functional illiteracy.
* Any contraindication to any test or procedure at the time of study inclusion.
* Family history of monogenic AD.
* Not willing to undergo one or more of the tests and procedures described in the protocol at baseline.

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Offsprings of subjects diagnosed of probable AD before reaching 75 years of age, according to McKhann et al. [McKhann et al., 1984] criteria, will be selected from spontaneous volunteers and Alzheimer's patients associations members.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from preclinical phase of AD to Mild Cognitive Impairment. | Every 3 years, from date of inclusion until the date of first documented progression, fulfilling mild cognitive impairment criteria, or date of death from any cause, whichever came first, assessed up to 12 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Molinuevo, MD, PhD, Principal Investigator — Scientific Director
Locations (1):
- Barcelonabeta Brain Research Center, Barcelona, Spain

REFERENCES:
- [Derived] Lazaro I, Brugulat-Serrat A, Suarez-Calvet M, Fauria K, Minguillon C, Gispert JD, Molinuevo JL, Harris WS, Sanchez-Benavides G, Grau-Rivera O, Sala-Vila A; ALFA study. Red blood cell omega-3 status and longitudinal cognition in individuals at risk of Alzheimer disease. J Nutr. 2025 Dec;155(12):4514-4522. doi: 10.1016/j.tjnut.2025.09.032. Epub 2025 Sep 27. PMID 41022152
- [Derived] Akinci M, Aguilar-Dominguez P, Palpatzis E, Shekari M, Garcia-Prat M, Deulofeu C, Fauria K, Garcia-Aymerich J, Gispert JD, Suarez-Calvet M, Grau-Rivera O, Sanchez-Benavides G, Arenaza-Urquijo EM; ALFA study. Physical activity changes during midlife link to brain integrity and amyloid burden. Alzheimers Dement. 2025 May;21(5):e70007. doi: 10.1002/alz.70007. PMID 40304268
- [Derived] Brugulat-Serrat A, Sanchez-Benavides G, Cacciaglia R, Salvado G, Shekari M, Collij LE, Buckley C, van Berckel BNM, Perissinotti A, Ninerola-Baizan A, Mila-Aloma M, Vilor-Tejedor N, Operto G, Falcon C, Grau-Rivera O, Arenaza-Urquijo EM, Minguillon C, Fauria K, Molinuevo JL, Suarez-Calvet M, Gispert JD; ALFA Study. APOE-epsilon4 modulates the association between regional amyloid deposition and cognitive performance in cognitively unimpaired middle-aged individuals. EJNMMI Res. 2023 Mar 1;13(1):18. doi: 10.1186/s13550-023-00967-6. PMID 36856866
- [Derived] Akinci M, Pena-Gomez C, Operto G, Fuentes-Julian S, Deulofeu C, Sanchez-Benavides G, Mila-Aloma M, Grau-Rivera O, Gramunt N, Navarro A, Minguillon C, Fauria K, Suridjan I, Kollmorgen G, Bayfield A, Blennow K, Zetterberg H, Molinuevo JL, Suarez-Calvet M, Gispert JD, Arenaza-Urquijo EM; ALFA Study. Prepandemic Alzheimer Disease Biomarkers and Anxious-Depressive Symptoms During the COVID-19 Confinement in Cognitively Unimpaired Adults. Neurology. 2022 Oct 4;99(14):e1486-e1498. doi: 10.1212/WNL.0000000000200948. Epub 2022 Aug 2. PMID 35918160
- [Derived] Mila-Aloma M, Brinkmalm A, Ashton NJ, Kvartsberg H, Shekari M, Operto G, Salvado G, Falcon C, Gispert JD, Vilor-Tejedor N, Arenaza-Urquijo EM, Grau-Rivera O, Sala-Vila A, Sanchez-Benavides G, Gonzalez-de-Echavarri JM, Minguillon C, Fauria K, Ninerola-Baizan A, Perissinotti A, Kollmorgen G, Suridjan I, Zetterberg H, Molinuevo JL, Blennow K, Suarez-Calvet M; ALFA Study. CSF Synaptic Biomarkers in the Preclinical Stage of Alzheimer Disease and Their Association With MRI and PET: A Cross-sectional Study. Neurology. 2021 Nov 23;97(21):e2065-e2078. doi: 10.1212/WNL.0000000000012853. Epub 2021 Sep 23. PMID 34556565
- [Derived] Mila-Aloma M, Shekari M, Salvado G, Gispert JD, Arenaza-Urquijo EM, Operto G, Falcon C, Vilor-Tejedor N, Grau-Rivera O, Sala-Vila A, Sanchez-Benavides G, Gonzalez-de-Echavarri JM, Minguillon C, Fauria K, Ninerola-Baizan A, Perissinotti A, Simon M, Kollmorgen G, Zetterberg H, Blennow K, Suarez-Calvet M, Molinuevo JL; ALFA study. Cognitively unimpaired individuals with a low burden of Abeta pathology have a distinct CSF biomarker profile. Alzheimers Res Ther. 2021 Jul 27;13(1):134. doi: 10.1186/s13195-021-00863-y. PMID 34315519
- [Derived] Grau-Rivera O, Navalpotro-Gomez I, Sanchez-Benavides G, Suarez-Calvet M, Mila-Aloma M, Arenaza-Urquijo EM, Salvado G, Sala-Vila A, Shekari M, Gonzalez-de-Echavarri JM, Minguillon C, Ninerola-Baizan A, Perissinotti A, Simon M, Kollmorgen G, Zetterberg H, Blennow K, Gispert JD, Molinuevo JL; ALFA Study. Association of weight change with cerebrospinal fluid biomarkers and amyloid positron emission tomography in preclinical Alzheimer's disease. Alzheimers Res Ther. 2021 Feb 17;13(1):46. doi: 10.1186/s13195-021-00781-z. PMID 33597012
- [Derived] Arenaza-Urquijo EM, Salvado G, Operto G, Minguillon C, Sanchez-Benavides G, Crous-Bou M, Grau-Rivera O, Sala-Vila A, Falcon C, Suarez-Calvet M, Zetterberg H, Blennow K, Gispert JD, Molinuevo JL; ALFA Study. Association of years to parent's sporadic onset and risk factors with neural integrity and Alzheimer biomarkers. Neurology. 2020 Oct 13;95(15):e2065-e2074. doi: 10.1212/WNL.0000000000010527. Epub 2020 Jul 31. PMID 32737076
- [Derived] Salvado G, Molinuevo JL, Brugulat-Serrat A, Falcon C, Grau-Rivera O, Suarez-Calvet M, Pavia J, Ninerola-Baizan A, Perissinotti A, Lomena F, Minguillon C, Fauria K, Zetterberg H, Blennow K, Gispert JD; Alzheimer's Disease Neuroimaging Initiative, for the ALFA Study. Centiloid cut-off values for optimal agreement between PET and CSF core AD biomarkers. Alzheimers Res Ther. 2019 Mar 21;11(1):27. doi: 10.1186/s13195-019-0478-z. PMID 30902090